CLINICAL TRIAL: NCT00817089
Title: Defining an Endopheneotype for Alcohol Treatment With Naltrexone
Brief Title: Understanding Treatment Response With Naltrexone Among White Alcoholics
Acronym: DEFINE II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, David Oslin, Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 806019
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-10

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Groups 1 and 3 get placebo in session 1 and placebo in session 2, Groups 2 and 4 get placebo in session 1 and naltrexone in session 2
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 Asn40 Placebo Placebo (Placebo Comparator): Each alcohol session preceded by pretreatment with placebo oral tablet
  Interventions: Drug: Placebo Oral Tablet
- Group 2 Asn40 Placebo Naltrexone (Active Comparator): The first alcohol session preceded by pretreatment with placebo oral tablet. The second alcohol session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Interventions: Drug: Placebo Oral Tablet; Drug: Naltrexone
- Group 3 Asp40 Placebo Placebo (Placebo Comparator): Each alcohol session preceded by pretreatment with placebo oral tablet
  Interventions: Drug: Placebo Oral Tablet
- Group 4 Asp40 Placebo Naltrexone (Active Comparator): The first alcohol session preceded by pretreatment with placebo oral tablet. The second alcohol session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Interventions: Drug: Placebo Oral Tablet; Drug: Naltrexone

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo pill
  Other Names: Placebo
Drug: Naltrexone — 50 mg of naltrexone prior to challenge session
  Arms: Group 2 Asn40 Placebo Naltrexone; Group 4 Asp40 Placebo Naltrexone

SUMMARY:
This is a study involving treatment for alcohol dependence among males of European or Asian decent. The ultimate aim of this line of investigation is to further establish a genetic link between alcohol dependence and treatment by defining an endophenotype associated with treatment response. The study consists of two inpatient alcohol challenge sessions with treatment using random assignment to either naltrexone or placebo.

DETAILED DESCRIPTION:
Despite the well-established efficacy of naltrexone, there are significant variations in individual responses to naltrexone. A critical question remains: under what circumstances and for which patients will naltrexone be most beneficial? Recent work at our center provides evidence that the mu-opioid receptor (OPRM1) gene polymorphism A118G (Asn40Asp) imparts a significant change in treatment response. We have shown that patients with Asn40 variant (absence of heavy drinking -73.9% v/s 49% response). To further consolidate our knowledge, we wish to test the relationship between A118G polymorphism and the subjective/objective measures to alcohol among alcoholics treated with naltrexone. This work is focused on subjects of European or Asian decent as the A118G polymorphism occurs in less than 1% of those of African decent.

Up to 40 subjects will be recruited. The subjects were admitted to the UPenn Translational Research Center and receive two alcohol challenge sessions after pretreatment with naltrexone or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males 21 years of age or older of European or Asian decent.
2. Has a current DSM IV diagnosis of alcohol dependence as determined by the Structural Clinical Interview for DSM IV (SCID-IV Mini).
3. Drank an average of 21 drinks/week in the 60 days prior to treatment and had at least 2 occasions of heavy drinking (5 or more drinks on a given day for men), as measured by the Timeline Followback (TLFB).
4. Has adequate vision, hearing, and ability to communicate to allow study participation.
5. Successfully completes detoxification as manifested by at least 48 consecutive hours of no self-reported alcohol use immediately prior to admission to the inpatient unit.
6. Has signed a witnessed informed consent
7. Scores below an 8 on the Clinical Inventory of Withdrawal for Alcohol (CIWA) prior to starting naltrexone/placebo; and 8) Can speak, print, and understand English.

Exclusion Criteria:

1. Meets DSM-IV criteria for dependence on any substance other than alcohol or nicotine in the last 6 months.
2. Tests positive on the urine drug screen for opioids, cocaine, or amphetamine at the screening visit (only 1 repeat test permitted).
3. Meets current or lifetime DSM-IV criteria for bipolar affective disorder, schizophrenia, or any psychotic disorder
4. The presence of unstable or serious medical illness, including history of stroke, seizure disorder, severe liver disease (AST or ALT > 5x normal at the time of randomization), or unstable cardiac disease
5. Has taken any psychotropic medications (including disulfiram) regularly within the last seven days prior to randomization (14 days for fluoxetine) or needs immediate treatment with a psychotropic medication (with the exception of detoxification medications or benadryl used sparingly for sleep)
6. Over age 64 and has evidence of severe cognitive impairment as evidenced by a Mini-mental status exam (MMSE) score <24
7. Has suicidal or homicidal ideation necessitating inpatient hospitalization
8. Has been abstinent more than 14 days prior to Phase 1
9. Is of African Descent
10. Meets current DSM-IV criteria for for major depression (non-substance induced), PTSD, or panic disorder.
11. Has significant hematological, pulmonary, endocrine, cardiovascular, renal, or gastrointestinal disease.

Ages: 21 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Oslin, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Asn40 Placebo Placebo: Asn40: Placebo, Placebo
  Each alcohol session preceded by pretreatment with placebo.
  Placebo: placebo pills
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 2: Asn40 Placebo Naltrexone: Asn40: Placebo, Naltrexone
  The first alcohol challenge session preceded by pretreatment with placebo. The second alcohol challenge session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Placebo: placebo pills
  naltrexone: 50 mg of naltrexone prior to challenge session
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 3: Asp40 Placebo Placebo: Asp40: Placebo, Placebo
  Each alcohol challenge session preceded by pretreatment with placebo.
  Placebo: placebo pills
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 4: Asp40 Placebo Naltrexone: Asp40: Placebo, Naltrexone
  The first alcohol challenge session preceded by pretreatment with placebo. The second challegne alcohol session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Placebo: placebo pills
  naltrexone: 50 mg of naltrexone prior to challenge session
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
Period: First Alcohol Challenge
Arm/Group | Group 1: Asn40 Placebo Placebo | Group 2: Asn40 Placebo Naltrexone | Group 3: Asp40 Placebo Placebo | Group 4: Asp40 Placebo Naltrexone
Started | 6 | 8 | 4 | 6
Completed | 6 | 8 | 4 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Period: Second Alcohol Challenge
Arm/Group | Group 1: Asn40 Placebo Placebo | Group 2: Asn40 Placebo Naltrexone | Group 3: Asp40 Placebo Placebo | Group 4: Asp40 Placebo Naltrexone
Started | 6 | 8 | 4 | 5
Completed | 6 | 7 | 4 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Asn40 Placebo Placebo: Asn40: Placebo, Placebo
  Each alcohol challenge session preceded by pretreatment with placebo
  Placebo: placebo pills
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 2: Asn40 Placebo Naltrexone: Asn40: Placebo, Naltrexone
  The first alcohol challenge session preceded by pretreatment with placebo. The second challegne alcohol session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Placebo: placebo pills
  naltrexone: 50 mg of naltrexone prior to challenge session
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 3: Asp40 Placebo Placebo: Asp40: Placebo, Placebo
  Each alcohol challenge session preceded by pretreatment with placebo
  Placebo: placebo pills
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 4: Asp40 Placebo Naltrexone: Asp40: Placebo, Naltrexone
  The first alcohol challenge session preceded by pretreatment with placebo. The second alcohol challenge session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Placebo: placebo pills
  naltrexone: 50 mg of naltrexone prior to challenge session
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Total: Total of all reporting groups
Arm/Group | Group 1: Asn40 Placebo Placebo | Group 2: Asn40 Placebo Naltrexone | Group 3: Asp40 Placebo Placebo | Group 4: Asp40 Placebo Naltrexone | Total
Number analyzed (Participants) | 6 | 8 | 4 | 6 | 24
Age, Customized [Count of Participants; unit: Participants]
  <21 years | 0 | 0 | 0 | 0 | 0
  Between 21 and 65 years | 6 | 8 | 4 | 6 | 24
  >65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 8 | 4 | 6 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 8 | 4 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Biphasic Alcohol Effects Scale:Total Mood
Description: Change from baseline to peak cortisol response, during the 2nd alcohol challenge session, subjective response as measured by Biphasic Alcohol Effects Scale: Total Mood.
  Biphasic Alcohol Effects Scale: Total Mood: minimum = 0, maximum = 106, higher scores indicate better outcomes.
Time Frame: during 2nd alcohol challenge session
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1: Asn40 Placebo Placebo: Asn40: Placebo, Placebo
  Each alcohol challenge session preceded by pretreatment with placebo.
  Placebo: placebo pills
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
Arm/Group | Group 1: Asn40 Placebo Placebo | Group 2: Asn40 Placebo Naltrexone | Group 3: Asp40 Placebo Placebo | Group 4: Asp40 Placebo Naltrexone
Number analyzed (Participants) | 6 | 7 | 4 | 5
units on a scale | 6.94 (9.53) | 3.57 (18.46) | 6.50 (4.04) | 3.20 (8.11)

2. Secondary Outcome: Adrenocorticotropic Hormone (ACTH) Levels
Description: Change from baseline to peak cortisol response during the 2nd alcohol challenge session, objective response as measured by Adrenocorticotropic hormone (ACTH).
Time Frame: during 2nd alcohol challenge session
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Group 1 Asn40 Placebo Placebo: Asn40: Placebo, Placebo
  Each alcohol challenge session preceded by pretreatment with placebo.
  Placebo: placebo pills
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 2 Asn40 Placebo Naltrexone: Asn40: Placebo, Naltrexone
  The first alcohol challegne session preceded by pretreatment with placebo. The second alcohol challenge session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Placebo: placebo pills
  Naltrexone: 50 mg of naltrexone prior to challenge session
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 3 Asp40 Placebo Placebo: Asp40: Placebo, Placebo Each alcohol challenge session preceded by pretreatment with placebo oral tablet
  Placebo Oral Tablet: Placebo pill
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 4 Asp40 Placebo Naltrexone: Asp40: Placebo, Naltrexone
  The first alcohol challenge session preceded by pretreatment with placebo oral tablet. The second alcohol challenge session preceded by pretreatment with naltrexone 50 mg as a single dose.
  Placebo Oral Tablet: Placebo pill
  Naltrexone: 50 mg of naltrexone prior to challenge session
  alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice
Arm/Group | Group 1 Asn40 Placebo Placebo | Group 2 Asn40 Placebo Naltrexone | Group 3 Asp40 Placebo Placebo | Group 4 Asp40 Placebo Naltrexone
Number analyzed (Participants) | 6 | 7 | 4 | 5
pg/ml | -7.83 (14.34) | 3.86 (7.47) | 5.25 (8.42) | -3.20 (14.10)

ADVERSE EVENTS:
Time Frame: 36 hours
Description: Adverse events were tracked in the 36 hours after the second alcohol challenge session
Groups:
- Group 1: Asn40 Placebo Placebo: Asn40: placebo, placebo
  Each alcohol challenge session preceded by pretreatment with placebo.
  placebo: placebo pills
  alcohol : 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 2: Asn40 Placebo Naltrexone: Asn40: placebo, naltrexone
  The first alcohol challenge session preceded by pretreatment with placebo. The second alcohol challenge session preceded by pretreatment with naltrexone 50 mg as a single dose.
  placebo: placebo pills
  naltrexone : 50 mg of naltrexone prior to challenge session
  alcohol : 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 3: Asp40 Placebo Placebo: Asp40: placebo, placebo prior
  Each alcohol challenge session preceded by pretreatment with placebo.
  placebo: placebo pills
  alcohol : 190 proof alcohol prepared to 11% volume mixed with fruit juice
- Group 4: Asp40 Placebo Naltrexone: Asp40: placebo, naltrexone
  The first alcohol challenge session preceded by pretreatment with placebo. The second alcohol challenge session preceded by pretreatment with naltrexone 50 mg as a single dose.
  placebo: placebo pills
  naltrexone : 50 mg of naltrexone prior to challenge session
  alcohol : 190 proof alcohol prepared to 11% volume mixed with fruit juice
Arm/Group | Group 1: Asn40 Placebo Placebo | Group 2: Asn40 Placebo Naltrexone | Group 3: Asp40 Placebo Placebo | Group 4: Asp40 Placebo Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/4 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No